CLINICAL TRIAL: NCT06790329
Title: Endoscopic Sleeve Gastroplasty With Fundal Mucosal Ablation - a Pilot Study
Brief Title: ESG With Fundal Mucosal Ablation
Acronym: ESG-FUMA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Stephen KK Ng, Principal Investigator, Chinese University of Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CRE-2024.501
Record Dates: First submitted 2025-01-17; First posted 2025-01-24 (Actual); Last update posted 2025-01-24 (Actual); Status verified 2025-01

CONDITIONS: Obesity and Obesity-related Medical Conditions
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Endoscopic sleeve gastroplasty with fundal mucosal ablation (Experimental): First part of procedure - endoscopic gastric fundus mucosal ablation Second part of procedure - endoscopic sleeve gastroplasty
  Interventions: Procedure: Endoscopic sleeve gastroplasty with fundal mucosal ablation

INTERVENTIONS:
Procedure: Endoscopic sleeve gastroplasty with fundal mucosal ablation — Mucosal ablation around the gastric fundus is initially performed using a hybrid argon plasma coagulation (H-APC) probe, following a submucosal saline injection, until ablation coagulum is visible. Subsequently, endoscopic sleeve gastroplasty (ESG) is performed using a full-thickness endoscopic suturing device (Overstitch, Apollo). This is done in a standard manner, employing 6-8 permanent full-thickness sutures along the greater curvature of the stomach in a running plication, starting from the angular incisura and extending proximally while sparing the fundus. Hemostasis is carefully checked and confirmed before the procedure is completed.

SUMMARY:
Endoscopic sleeve gastroplasty (ESG) have emerged as an effective primary endoscopic therapy for weight loss. While ESG recapitulates the configuration of a gastric sleeve, it has not yet been shown to achieve as robust weight loss outcomes compared to the laparoscopic sleeve gastrectomy (LSG). A major difference between ESG and LSG is that the former does not involve the gastric fundus and therefore does not lead to decrease in fasting plasma ghrelin after procedure.

Recently, a new endoscopic technique involving the ablation of the gastric fundus has been developed, showing promising results with a reduction in fasting plasma ghrelin levels and a mean total body weight loss of 7.7%. Combining endoscopic gastric fundus mucosal ablation with ESG could potentially enhance the weight loss effects of ESG while maintaining an acceptable safety profile.

This pilot study aims to evaluate the efficacy, safety, and physiological effects of combining endoscopic sleeve gastroplasty with fundal mucosal ablation (ESG-FUMA) in obese patients eligible for endoscopic bariatric therapies.

ELIGIBILITY:
Inclusion Criteria:

* BMI equal or more than 30kg/m2 (27.5kg/m2 for Chinese or South Asian) to 40kg/m2, or BMI equal or more than 40kg/m2 and patient is either high risk for surgery or unwilling to undergo surgery, AND
* failed standard obesity therapy of diet, exercise, behavior modification, and pharmacologic agents either alone or in combination

Exclusion Criteria:

* Previous upper GI surgery (e.g. bariatric surgery, anti-reflux surgery; gastrectomy; esophageal surgery)
* Previous ESG
* Gastroparesis
* Active smoking
* An ongoing or a history of treatment with opioids in the last 12 months prior to enrollment
* Previous pyloromyotomy or pyloroplasty
* Gastrointestinal obstruction
* Use of any medication that may interfere with weight loss or gastric emptying
* Severe coagulopathy
* Esophageal or gastric varices and/or portal hypertensive gastropathy
* Underlying uncontrolled endocrine problem that leads to obesity. (e.g. Hypothyroidism, Cushing syndrome, eating disorder etc.)
* Any inflammatory disease of the gastrointestinal tract (including but not limited to severe (LA Grade C or D) esophagitis, active gastric ulceration, active duodenal ulceration, or specific inflammation such as Crohn's disease)
* Malignancy
* Pregnant or breast feeding
* Patients not fit for general anesthesia
* ASA grade IV or V
* Mental or psychiatric disorder; Drug or alcohol addiction
* Other cases deemed by the examining physician as unsuitable for safe treatment
* Refusal to participate

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Body weight | baseline, 1,3,6,12 months
  Weight change compared to baseline

SECONDARY OUTCOMES:
Adverse events | within 30 days of procedure
  Adverse events relating to endoscopic intervention, graded according to the Common Terminology Criteria for Adverse Events (CTCAE)
Technical success rate | 1 day
  successful completion of endoscopic procedures
Serum ghrelin levels | baseline, 3,6,12 months
  Serum ghrelin levels compared to baseline
Blood pressure | baseline, 1,3,6,12 months
  Blood pressure and anti-hypertensive medication use compared to baseline
Lipid profile | baseline, 3,6,12 months
  Lipid profile compared to baseline
Pain scale after procedure | 3 days
  measured by visual analogue scale (0:no pain - 10:worst pain)
Change in Quality of Life | baseline, 3,6,12 months
  measured by 36-Item Short Form Survey (SF-36) questionnaire - (score 0:worst - 100:best)
Gastric emptying symptoms | baseline, 3,6,12 months
  measured by gastroparesis cardinal symptom index (GCSI) - (0:best - 45:worst)
Eating behaviors | baseline, 3,6,12 months
  measured by Three-Factor Eating Questionnaire (TFEQ-R21) - (21:worst - 84:best)
Fasting glucose level | baseline, 3,6,12 months
  levels compared to baseline
Insulin level | baseline, 3,6,12 months
  levels compared to baseline
HbA1c level | baseline, 3,6,12 months
  levels compared to baseline
hepatic steatosis index | baseline, 3,6,12 months
  level compared to baseline
NAFLD fibrosis | baseline, 3,6,12 months
  NAFLD fibrosis scores compared to baseline (F0: no liver fibrosis - F4: significant liver fibrosis)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Ng, FRCSEd(Gen), Principal Investigator — Prince of Wales Hospital, the Chinese University of Hong Kong
Locations (1):
- Chinese University of Hong Kong, Shatin, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided